CLINICAL TRIAL: NCT06503614
Title: ENHANCE (Elevated NKG2A and HLA-E Amplify NK/CD8 Checkpoint Engagers): A Phase 2 Trial of Durvalumab (MEDI4736) Plus Monalizumab in Non-Muscle-Invasive Bladder Cancer
Brief Title: A Trial of Durvalumab (MEDI4736) Plus Monalizumab in Non-Muscle-Invasive Bladder Cancer
Acronym: ENHANCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Sfakianos (Other)
Collaborators: AstraZeneca (Industry); Icahn School of Medicine at Mount Sinai (Other); Bladder Cancer Advocacy Network (Other)
Responsible Party: Sponsor-Investigator, John Sfakianos, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU21-551
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle Invasive Bladder Cancer; Non-Muscle Invasive Bladder Urothelial Carcinoma
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — durvalumab; monalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Durvalumab and Monalizumab for CIS +/- high grade papillary urothelial cancer (Experimental): Durvalumab 1500mg IV and monalizumab 1500mg IV will be administered to all patients once every 4 weeks. A cycle is equal to 4 weeks. This will continue until disease progression, unacceptable toxicity, or for a maximum of 1 year.
  Interventions: Drug: Durvalumab; Drug: Monalizumab
- Cohort B: Durvalumab and Monalizumab for high grade papillary urothelial cancer without CIS (Experimental): Durvalumab 1500mg IV and monalizumab 1500mg IV will be administered to all patients once every 4 weeks. A cycle is equal to 4 weeks. This will continue until disease progression, unacceptable toxicity, or for a maximum of 1 year.
  Interventions: Drug: Durvalumab; Drug: Monalizumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg IV
  Other Names: MEDI 4736
Drug: Monalizumab — Monalizumab 1500mg IV

SUMMARY:
This is a phase 2 open-label two cohort study of durvalumab plus monalizumab in patients with BCG-unresponsive or BCG-exposed CIS NMIBC. Arm A will enroll 43 participants who have cancer in situ (CIS) with or without high grade papillary urothelial cancer. Arm B will enroll 17 participants who do not have cancer in situ (CIS) but do have high grade papillary urothelial cancer. Eligible patients will be enrolled to receive up to 13 cycles of monthly combination of monalizumab and durvalumab. Both monalizumab and durvalumab will be administered intravenously (IV) every 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of consent.
2. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up. Able and willing to provide written informed consent.
3. Eastern Cooperative Oncology Group scores ≤ 1 within 28 days prior to registration.
4. Non-muscle-invasive bladder cancer

   * Cohort A: CIS +/- high grade papillary urothelial cancer (Ta or T1) after 3-mo evaluation after induction BCG.
   * Cohort B: High grade papillary urothelial cancer (Ta or T1) after 3-mo evaluation after induction BCG.
5. Mixed variant histology (adenocarcinoma, squamous cell carcinoma) is eligible, but pure variant histology is ineligible. NOTE: Pathology report required for documentation purposes.
6. Patients can have BCG-unresponsive or BCG-exposed NMIBC11. Adequate BCG therapy is defined as completing at least induction BCG (≥ 5 doses) and the first round of maintenance or second induction course BCG (≥ 2 doses). The subsequent round of BCG, either maintenance or repeat induction, must be given within 6 months of initial induction BCG.

   * BCG-unresponsive is defined as high grade persistent or recurrent NMIBC that has not achieved a disease-free status after an adequate course of BCG therapy. This includes patients with:

     * Persistent or recurrent high-grade tumors (Ta/T1) or carcinoma in situ (CIS) within 6 to 12 months of completing adequate BCG therapy.
     * Recurrent high-grade papillary disease within 6 months of BCG therapy.
     * High-grade T1 disease found at the first evaluation after BCG induction therapy alone.
   * BCG-exposed is defined as high grade NMIBC that has recurred after an initial response or is still present after initial treatment, but recurrence is never too late to be considered "BCG-unresponsive". This includes patients with:

     * High-grade recurrence between 12 and 24 months after adequate BCG therapy.
     * Recurrence within 24 months of inadequate BCG therapy.
     * High-risk recurrence at the 3-month mark after an initial BCG induction.
     * High grade recurrence (T1, Ta, CIS) while on maintenance therapy would be eligible. The recurrence must be within 6 months of the last BCG dose.
7. Patients may have received up to 2 lines of prior therapy (including chemotherapy or other approved agents) for NMIBC (NOTE: prior PD-1/PD-L1 blockade is prohibited).
8. Patients must be deemed unfit for radical cystectomy by the treating physician or refuse radical cystectomy. NOTE: Reason for being deemed unfit or refusal should be documented in the medical record.
9. All visible tumor must be completely resected within 60 days prior to registration (residual pure CIS is permitted).

   * All patients must have had a cystoscopy (or TURBT with complete resection) without papillary tumor and negative urine cytology within 28 days prior to registration (positive cytology is allowed in patients with CIS).
10. All patients with T1 tumors must undergo restaging TURBT within 60 days prior to registration.

    * There must be uninvolved muscularis propria in the restaging TURBT specimen.
    * The initial TURBT prior to the restaging TURBT may be > 60 days prior to registration.
11. Patients must have baseline tumor tissue from either initial or repeat TURBTs for submission of a minimum of 2 and up to 10 unstained slides for translational study objectives. If archival tissue is not available, the subject is not eligible.
12. Adequate organ function as defined by ALL of the following within 28 days prior to registration:

    * Absolute neutrophil count ≥ 1500/µL
    * Platelets ≥ 100,000/µL
    * Hemoglobin ≥ 9 g/dL
    * Aspartate aminotransferase/alanine aminotransferase ≤ 1.5× upper limit of normal (ULN)
    * Total serum bilirubin ≤ 1.5×ULN*; *Patients with Gilbert's disease: ≤ 3×ULN
    * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5×ULN unless the patient is on therapeutic anticoagulation.
    * Creatinine clearance ≥ 40 mL/min by Cockcroft-Gault estimation. The patient's estimated CrCl will be calculated by the local laboratory (for eligibility purposes) using screening/baseline height (m), actual weight (kg), and serum creatinine:

    Males: CrCl = ((140 - age in years) × weight (kg)) / (72× serum creatinine (mg/dL)) Females: CrCl = ((140 - age in years) × weight (kg) ×0.85) / (72× serum creatinine (mg/dL))
13. Females of childbearing potential (FOCBP) must have a negative urine or serum pregnancy test within 7 days of registration. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required. FOCBP must agree to use contraception during the study.
14. Men capable of fathering a child must agree to use contraception during the study.
15. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
2. Prior CIS of the ureters or prostatic urethra within 24 months prior to registration.
3. Evidence of metastatic disease on imaging (CT or MRI) of the abdomen and pelvis within 90 days of registration.
4. Body weight ≤ 30 kg.
5. History of allogeneic organ transplantation.
6. History of another primary malignancy other than muscle-invasive bladder cancer less than 5 years prior to Day 1 of this trial, with the exception of a malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study drug and of low potential risk for recurrence. Other exceptions include those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer (non-melanoma skin cancer) or lentigo maligna without evidence of disease, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ without evidence of disease treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate specific antigen [PSA] ≤ 10 mg/mL, etc.)
7. Currently participating in or has participated in a trial of an investigational agent within 4 weeks prior to the first dose of study treatment or 5 half-lives, whichever is longer without recovery of clinically significant toxicities from that therapy.
8. Active or prior autoimmune or inflammatory disorders requiring systemic treatment within 24 months prior to registration. Autoimmune or inflammatory disorders include, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease(colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis),antiphospholipid syndrome, Sarcoidosis syndrome, or Wegener's syndrome (granulomatosis with polyangiitis, Graves' disease, hypophysitis, uveitis, etc), Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. NOTE: The following are exceptions to this criterion: Patients with vitiligo or alopecia, hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement. Any chronic skin condition that does not require systemic therapy. Patients without active disease in the last 5 years may be included but only after consultation with the study physician. Patients with celiac disease controlled by diet alone.
9. A diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to registration. NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
10. Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
11. Active known tuberculosis.
12. Symptomatic herpes zoster within the past 30 days.
13. Active infection requiring systemic therapy. NOTE: Prophylactic antibiotics are permitted. Treatment for a UTI is allowed but must be deemed adequately treated by the treating physician prior the start of C1D1.
14. History of idiopathic pulmonary fibrosis or organizing pneumonia.
15. History of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
16. Patients known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) are eligible with the following:

    * On effective anti-retroviral therapy with undetectable viral load within 6 months of registration.
    * HIV-infected participants must not have a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
17. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. NOTE: No testing for Hepatitis B and Hepatitis C is required unless mandated by a local health authority.
18. Participants with a known co-infection with HBV and HCV, or co-infection with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti HBcAb with detectable HBV DNA); AND HCV positive (presence of anti-HCV antibodies); OR HDV positive (presence of anti-HDV antibodies).
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Received live vaccines within 30 days of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. COVID-19 vaccinations are permitted.
21. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study drug. Note: Local surgery of isolated lesions for palliative intent is acceptable.
22. Uncontrolled intercurrent illness, including but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
23. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
24. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control.
25. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
26. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
27. History of leptomeningeal carcinomatosis
28. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
29. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 6 months
  Complete response will be determined by bladder biopsy and urinary cytology for malignancy for subjects with a CIS component at 6 months CT/MRI urography will be used to rule out extravesical disease. (Cohort A)

SECONDARY OUTCOMES:
Incidence of treatment related Adverse Events | 12 months
  Safety will be determined by summarizing all treatment related adverse events according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5. (Cohort A and B)
Progression-free Survival (PFS) | 36 months
  Progression-free survival (PFS) will be measured from the date of study registration to the date of progression or death due to any cause, whichever occurs first. Surviving patients without any documented progression will be censored at the date of last known contact. Progression will be defined as the development of muscle invasive bladder cancer or metastatic urothelial cancer (nodal and/or distant). (Cohort A)
Overall Survival (OS) | 36 months
  Overall survival (OS) will be measured from the date of study registration to date of death due to any cause. Surviving patients will be censored at the date of last known contact. (Cohort A)
Event Free Survival | 36 months
  Event-free survival will be measured from the date of study registration to the first documentation of an event. Patients without documented events and who are still alive, will be censored at last disease assessment. Patients who start any subsequent anti- cancer therapy without any reported events will be censored at their last disease assessment. (Cohort A)
Cyctectomy Free Survival | 36 months
  Cystectomy-free survival will be measured from the date of study registration to the date of cystectomy for all patients. (Cohort A)
Duration of Response (DOR) | 36 months
  Duration of response (DOR) will be measured from the time a patient had a documented response (the time would start at the time a response was first noted) until disease-progression. This analysis will only include those patients in the CIS population who achieve a response. Patients who are alive and without a documented progression at the time of analysis will be censored at the time of the last disease status evaluation. (Cohort A)
Recurrence-free Survival | 12 months
  Recurrence-free survival will be measured from the date of study registration to the date of recurrence. Recurrence will be defined as the development of high-grade bladder cancer for patients without a CIS component at baseline. (Cohort B)

CONTACTS AND LOCATIONS:
Overall Officials: John Sfakianos, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York